CLINICAL TRIAL: NCT07378475
Title: Evaluation of the Effectiveness of Manual Lymphatic Drainage in Young Women With Primary Dysmenorrhea
Acronym: EDLMDP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Camilo Jose Cela University (Other)
Responsible Party: Principal Investigator, Edurne Úbeda D'Ocasar, Doctor, Camilo Jose Cela University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCJCDLMDP
Record Dates: First submitted 2025-12-20; First posted 2026-01-30 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Dysmenorrhea Primary
Keywords: Manual Lymphatic Drainage; physiotherapy
MeSH Terms: interventions — Manual Lymphatic Drainage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Manual Lymphatic Drainage Group (Experimental): All enrolled participants (N=20) will receive the intervention consisting of manual lymphatic drainage (MLD) following the Vodder method. The treatment will be applied during the late luteal phase (5-7 days before menstruation) in three consecutive menstrual cycles. Each session will last approximately 30-45 minutes and will include preparatory maneuvers (terminus, solar plexus, inguinal chains) and abdominal drainage sequence. No control group is included in this pilot study.
  Interventions: Other: Manual Lymphatic Drainage (MLD)

INTERVENTIONS:
Other: Manual Lymphatic Drainage (MLD) — This method, part of complex decongestive physiotherapy, involves gentle massage techniques that stimulate lymphatic circulation and venous return. Participants will receive three sessions of MLD during the late luteal phase (5-7 days before menstruation) over three consecutive menstrual cycles. Each session will last approximately 30-45 minutes and will follow the Vodder method, including preparatory maneuvers (terminus, solar plexus, inguinal chains) and abdominal drainage sequence.
  Frequency: One session per cycle for three months.

SUMMARY:
This pilot clinical trial aims to evaluate the effectiveness of manual lymphatic drainage (MLD) in reducing symptoms associated with primary dysmenorrhea in young women. Primary dysmenorrhea is a common gynecological condition characterized by intense pelvic pain during menstruation, often accompanied by fatigue, headache, and sleep disturbances. Despite its high prevalence, it is frequently underestimated, negatively impacting quality of life and daily activities.

The intervention consists of three monthly sessions of MLD performed during the late luteal phase, prior to menstruation. Outcome measures include pain intensity, abdominal circumference, pressure pain threshold, sleep quality, and health-related quality of life.

DETAILED DESCRIPTION:
Primary dysmenorrhea (PD) is defined as menstrual pain of uterine origin occurring in the absence of pelvic pathology. It typically affects adolescents and young women with regular ovulatory cycles. The pathophysiology involves hormonal changes during the late luteal phase, leading to increased prostaglandin synthesis, uterine hypercontractility, ischemia, and heightened nociceptive sensitivity.

Non-pharmacological interventions such as physical therapy techniques have shown promising results in alleviating symptoms. Manual lymphatic drainage (MLD), based on the Vodder method, uses gentle, rhythmic maneuvers to stimulate lymphatic flow, reduce tissue congestion, and promote parasympathetic activation, potentially improving pain perception and associated symptoms.

This study will assess whether MLD reduces pain intensity, abdominal swelling, and improves sleep quality and overall quality of life in women with PD.

ELIGIBILITY:
Inclusion Criteria:

* Female participants aged 18-25 years
* Confirmed diagnosis of primary dysmenorrhea
* Regular menstrual cycles
* Ability to provide informed consent

Exclusion Criteria:

* Secondary dysmenorrhea
* Use of hormonal contraceptives
* Presence of pelvic pathology (endometriosis, polycystic ovary syndrome, fibroids)
* Irritable bowel syndrome
* Use of analgesics or anti-inflammatory drugs within 12 hours prior to intervention
* Any therapy for dysmenorrhea in the previous month
* Pregnancy or suspected pregnancy
* Irregular menstrual cycles

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-01-30 (Estimated); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
VAS | baseline assessment, in the menstrual assessment of the first, second, and third months, and in the follow-up (fourth month)
  Change in pain intensity measured by Visual Analog Scale (VAS). Visual Analog Scale (0-10 cm) to assess menstrual pain intensity. Scores are classified as mild dysmenorrhoea (1-3 points), moderate dysmenorrhoea (4-7 points) and severe dysmenorrhoea (8-10 points).

SECONDARY OUTCOMES:
Pressure Pain Threshold (Algometry) | pre and post-intervention measurement in first month, pre and post-intervention measurement in the second month, pre and postintervention measurement in the third month, and in forth month (follow up)
  Measured bilaterally at L2 and S2 esclerotomes using a Fischer algometer (FPK-20). The tests will be carried out in the late luteal phase.
Abdominal Circumference (Circumferential Measurement) | second day of menstruation in the first month (baseline), second day of menstruation in the second month, second day of menstruation in the third month, and second day of menstruation in the fourth month (follow-up)
  Measured at supraumbilical and infraumbilical levels using a flexible tape.
Pittsburgh Sleep Quality Index questionnaire. | baseline assessment, post intervention in third month, and fourth month (follow-up)
  The Pittsburgh Sleep Quality Index (PSQI) was used to assess sleep quality, which allows the impact of menstrual pain on rest to be determined.The total score ranges from 0 to 21, where values greater than 5 indicate poor quality and values equal to or less than 5 reflect adequate rest.
Health-Related Quality of Life (EQ-5D-5L) | baseline assessment, post intervention in third month, and fourth month (follow-up)
  EuroQol questionnaire assessing mobility, self-care, usual activities, pain/discomfort, and anxiety/depression.This scale ranges from 0 to 100, with 0 being the worst possible health status and 100 being the best health status.
Dysmenorrhea Severity (WaLIDD Score) | baseline assessment, post intervention in third month, and fourth month (follow-up)
  Validated tool assessing work ability, pain location, intensity, and duration. The severity level is classified as: no dysmenorrhea (0), mild (1-4), moderate (5-7), and severe (8-12).
Andersh and Milsom dysmenorrhoea scale | baseline assessment, post intervention in third month, and fourth month (follow-up)
  The severity of dysmenorrhoea will be assessed using the Andersch and Milsom Scale, which classifies pain into four grades (0-3): grade 0 (no pain or limitation), grade 1 (mild pain with minimal interference), grade 2 (moderate pain with some interference with activities and relief with analgesics) and grade 3 (severe pain with marked limitation and poor response to treatment).
Menstrual Symptom Questionnaire (MSQ) | baseline assessment, post intervention in third month, and fourth month (follow-up)
  The Menstrual Symptom Questionnaire (MSQ) allows two forms of dysmenorrhoea to be assessed: spasmodic and congestive. The first 24 items assess symptoms characteristic of each type, with responses on a scale from 1 ('never') to 5 ('always'). Items associated with spasmodic dysmenorrhoea (S) are scored directly, while those associated with congestive dysmenorrhoea (C) are scored inversely. The final item (25) allows the participant to identify the type of dysmenorrhoea that best describes her experience. The total score ranges from 29 to 125 points, with higher values reflecting greater intensity of menstrual symptoms.

OTHER OUTCOMES:
Age | baseline
  Age (years)
Characteristics of dysmenorrhoea. Regularity | baseline
  Regularity of the menstrual cycle
Characteristics of dysmenorrhoea. Menarche | baseline
  Age at menarche
Characteristics of dysmenorrhoea. Duration. | baseline
  Duration of menstruation.
Characteristics of dysmenorrhoea. History. | baseline
  gynaecological history and use of cycle-related medication (contraceptives, analgesics, anti-inflammatories) or other medical indications.
Weight | baseline
  weight, measured in kilograms
BMI | baseline
  body mass index

CONTACTS AND LOCATIONS:
Overall Officials: Edurne Úbeda Docasar, Doctor, Principal Investigator — University Camilo José Cela